CLINICAL TRIAL: NCT04341350
Title: Comparison of an Inhaled Sedation Strategy to an Intravenous Sedation Strategy in Intensive Care Unit Patients Treated With Invasive Mechanical Ventilation : INASED Study
Brief Title: Comparison of an Inhaled Sedation Strategy to an Intravenous Sedation Strategy in Intensive Care Unit Patients Treated With Invasive Mechanical Ventilation
Acronym: INASED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INASED (29BRC19.0280)
Record Dates: First submitted 2020-03-09; First posted 2020-04-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Prevention of Delirium
MeSH Terms: interventions — Propofol; Acetaminophen; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual sedation (Active Comparator): Sedation according to a written, standardized Nurse management protocol using at least one sedative drug (propofol) and one analgesic drug.
  Interventions: Drug: Propofol + analgesic drug
- Inhaled sedation (Experimental): Sedation by inhalation of halogenated gas (Isoflurane) delivered by the Anesthetic-Conserving Device (ACD) system ANACONDA ™ associated with the administration of an analgesic drug.
  Interventions: Drug: Isoflurane + analgesic drug

INTERVENTIONS:
Drug: Propofol + analgesic drug — sedation according to a written, standardized Nurse management protocol using at least one sedative drug (propofol) and one analgesic drug. It uses the nurse driven analgesia protocol of each ward involved in the study. It uses a pain assessment score (BPS, VICOMORE, FLACC), local or regional anesthesia, non-opioïd adjuncts (acetaminophen, NSAIDs, nefopam), opioïds (per os opioïds, bolus of sufentanyl followed by continuous infusion if necessary, continuous infusion of remifentanyl
  Arms: Usual sedation
Drug: Isoflurane + analgesic drug — sedation by inhalation of halogenated gas (Isoflurane) delivered by the Anesthetic-Conserving Device (ACD) system ANACONDA ™ associated with the administration of a analgesic drug. It uses the nurse driven analgesia protocol of each ward involved in the study. It uses a pain assessment score (BPS, VICOMORE, FLACC), local or regional anesthesia, non-opioïd adjuncts (acetaminophen, NSAIDs, nefopam), opioïds (per os opioïds, bolus of sufentanyl followed by continuous infusion if necessary, continuous infusion of remifentanyl.
  Arms: Inhaled sedation

SUMMARY:
The objective of the study is to determine the impact on the frequency of occurrence of delirium of an early inhaled sedation strategy (from induction in rapid sequence if intubation in intensive care, or from admission if intubated in pre -hospital) by Isoflurane using an ANACONDA ™ type system, compared to a conventional intravenous sedation strategy.

DETAILED DESCRIPTION:
Sedation-analgesia is used in most patients treated with mechanical ventilation (MV). The usual benzodiazepine and morphine sedation reduces pain and anxiety and allows tolerance of invasive procedures in intensive care. These molecules, used as part of the sedation titration protocol or the daily sedation stop protocol, have improved patient outcomes.

Although necessary, these drugs, by mechanisms still uncertain, would promote the occurrence of resuscitation delirium. Delirium itself responsible for worsening morbidity and mortality (increase in the duration of MV, increase in the length of hospital stay, discussed increase in mortality, long-term cognitive sequelae).

This finding favored the use of new drugs in the sedation strategies of patients on MV. Dexmedetomidine has for example reduced the number of days of delirium, the number of days of coma and even mortality in septic patients. Its large-scale use has however been questioned by a recent study.

Halogenated gases have been used for a long time in anesthesia. Their pharmacodynamics, their positive and adverse effects, their therapeutic margins are well known. Thanks to technical innovations they can be used on resuscitation respirators. Several studies on targeted populations have shown the feasibility and the benefits of this use, in particular, the absence of accumulation, the absence of tachyphylaxis, the broad therapeutic range, the small interindividual variation, the rapidity of efficacy and the speed of awakening. Safety in use for the staff in charge of the patient is established. In addition, their potential neuroprotective effect would make it an anesthetic of choice in the prevention of resuscitation delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over
* Patient requiring mechanical ventilation for at least 24 hours
* The patient requires continuous and immediate sedation for more comfort, safety and to facilitate the administration of survival measures.
* Consent obtained from patient or relative

Exclusion Criteria:

Patient hospitalized for the following reasons for admission:

* Cardiac arrest
* State of refractory epilepticus
* Head trauma
* Stroke

  * Hearing, visual or aphasia disorders before inclusion making it impossible to take the CAM-ICU
  * Sedation started more than 24 hours ago
  * Impairment of cognitive functions and / or dementia
  * Contraindication to halogenated gases (personal or family history of malignant hyperthermia, acute or chronic neuromuscular disease, hepatocellular insufficiency with PT <30%)
  * Severe acute respiratory distress syndrome (ARDS) (Berlin criteria: PaO2 / FiO2 <100 after ventilatory optimisation))
  * PaCO2 at inclusion> 50 mmHg after ventilatory optimisation
  * Patient for whom a procedure of "limitation of active therapies" is envisaged at inclusion
  * Patient under guardianship or curatorship
  * Minor patient
  * Pregnant or breastfeeding woman
  * Patient not affiliated to the social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a delirium in intensive care | 28 days
  Occurrence of delirium in intensive care will be observed (yes / no)

SECONDARY OUTCOMES:
Mortality in intensive care | Throuh exit from the intensive care unit, an average of 28 days
  Mortality in intensive care will be observed
Mortality at day 28 | 28 days
  Mortality at day 28 will be observed
Hospital cost per patient | Through study completion, an average of 1 year.
  The average cost of hospitalization for each patient will be calculated taking into account their length of hospital stay, examinations carried out and medical treatment taken.
Number of days with vasopressors or inotropic agents | Throuh exit from the intensive care unit, an average of 28 days
  Number of days with vasopressors or inotropic agents will be observed
Number of days with sedation | Throuh exit from the intensive care unit, an average of 28 days
  Number of days with sedation will be observed
Cumulative dose anesthetics drugs | Throuh exit from the intensive care unit, an average of 28 days
  Cumulative dose anesthetics drugs will be observed
Duration of anesthetics drugs | Throuh exit from the intensive care unit, an average of 28 days
  Duration of anesthetics drugs will be observed
Maximum dose of vasopressors or inotropic agents | Throuh exit from the intensive care unit, an average of 28 days
  Maximum dose of vasopressors or inotropic agents will be observed
Ventilation free days at 28 days following randomisation | 28 days
  Ventilation free days at 28 days following randomisation will be observed
Incidence of delirium | 28 days
  Incidence of delirium will be observed
Duration of delirium | 28 days
  Duration of delirium will be observed
Length of ICU stay | Throuh exit from the intensive care unit, an average of 28 days
  Length of ICU stay will be calculated
Requirement of patients physical restraints | Throuh exit from the intensive care unit, an average of 28 days
  Requirement of physical restraints, of patients with unplanned extubation, unplanned catheter, urinary probe or gastric probe removal will be observed
Self aggressive act | Throuh exit from the intensive care unit, an average of 28 days
  Self aggressive act will be observed
Hetero-aggressive act | Throuh exit from the intensive care unit, an average of 28 days
  Hetero-aggressive act will be observed
Evaluation of cognitive functions | Through study completion, an average of 1 year.
  Cognitive function will be evaluated at discharge, 3- and 12 months using two kinds of score :
  * Cantab test, combining 6 cognitive evaluations with an iPad during a 45-60 minutes medical consultation
  * PCLS (Posttraumatic stress disorder Checklist Scale), HADS (Hospital Anxiety and Depression scale), SF36 (medical outcome study short form 36), IADL (instrumental activities of daily living) practised by a clinical research associate

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Bailly, MD, Principal Investigator — CHRU Brest
Locations (12):
- France (12):
  - CH Bourges, Bourges
  - CHU de Brest, Brest
  - CH Corbeil Essonnes, Corbeil-Essonnes
  - CH Le Mans, Le Mans
  - GHBS Lorient, Lorient
  - CH Melun, Melun
  - CHU Montpellier, Montpellier
  - CH Morlaix, Morlaix
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Tours - Réanimation Chirurgicale, Tours
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Bailly P, Egreteau PY, Ehrmann S, Thille AW, Guitton C, Grillet G, Reizine F, Huet O, Jaber S, Nowak E, L'her E. Inased (inhaled sedation in ICU) trial protocol: a multicentre randomised open-label trial. BMJ Open. 2021 Feb 19;11(2):e042284. doi: 10.1136/bmjopen-2020-042284. PMID 33608400